CLINICAL TRIAL: NCT04483336
Title: Effect of Virtual Reality Distraction on Pain and Anxiety During Infiltration Anesthesia in Pediatric Patients: A Randomized Clinical Trial
Brief Title: Virtual Reality Distraction During Dental Local Anesthesia Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Osama M Felemban, Assistant Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07072020
Record Dates: First submitted 2020-07-08; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Dental Anxiety; Dental Fear
Keywords: Dental Anxiety; Dental Fear; Infiltration Dental Local Anesthesia; Virtual Reality; Dental Pain
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Intervention Model Description: Subjects receiving dental local anesthesia were randomly assigned to wear VR goggles or watch a cartoon video on a regular screen.
Who Masked: Investigator
Masking Description: During the local anesthesia by the care provider, subjects in the test group had to wear VR goggles while control subjects watched a cartoon video on a TV screen. The pain and anxiety outcomes were assessed during the local anesthesia administration. Due to the nature of the study, it was not possible to mask the participants, care provider, or the outcome assessor. The investigator who statistically analyzed the data but was not involved in the dental procedures was masked to the group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality Distraction. (Experimental): Subjects watched a video cartoon using virtual reality goggles as a distraction technique during the administration of local anesthesia.
  Interventions: Other: Virtual Reality Distraction
- TV screen Distraction (Active Comparator): Subjects watched a video cartoon on a regular TV screen as a distraction technique during the administration of local anesthesia.
  Interventions: Other: TV Screen Distraction

INTERVENTIONS:
Other: Virtual Reality Distraction — Virtual reality goggles are commercially available wearable devices that are used to view view videos and play video games three dimensionally.
  Other Names: LG 360 virtual reality [VR] headset, LG Electronics
  Arms: Virtual reality Distraction.
Other: TV Screen Distraction — A cartoon video was played on a regular TV screen.
  Arms: TV screen Distraction

SUMMARY:
To evaluate the effect of virtual reality (VR) distraction on anxiety and pain during buccal infiltration anesthesia (BIA) in pediatric patients.

DETAILED DESCRIPTION:
Design and Participants: This randomized clinical trial was conducted including healthy, and cooperative 6-12-year-old children, with no known allergy and/or sensitivity to local anesthesia who are currently in need of nonemergency dental treatment under local anesthetic infiltration by one of the postgraduate or interns at the pediatric dentistry students, were eligible for the study. Patients with history of epilepsy and anxiety disorder were excluded from the study

Methods and Material: In the test group, subjects received BIA while being distracted using VR goggles; in the control group, subjects watched a cartoon video on a regular screen. Subjects' heart rate (HR) was measured at baseline and at four different timepoints during BIA administration to assess anxiety. The face, legs, activity, cry, consolability (FLACC) Behavioral Pain Assessment Scale was scored by two calibrated investigators to assess pain. After BIA, subjects rated their pain using the Arabic version of Wong-Baker FACES Pain Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 6-12-year-old children
* Cooperative during dental treatments
* In need of nonemergency dental treatment under local anesthetic infiltration

Exclusion Criteria:

* Allergy and/or sensitivity to local anesthesia
* Epilepsy
* Anxiety Disorder

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Dental Pain measured using the Wong-Baker FACES Pain Rating Scale | Immediately after the local anesthesia administration, subjects were put in an upright position and asked to rate their pain using a validated Arabic version of Wong-Baker FACES Pain Rating Scale.
  Wong-Baker FACES Pain Rating Scale is a six point scale (0, 2, 4, 6, 8, 10) where higher scores indicate worse pain.
Dental Pain and Behavior measured using Face, Legs, Activity, Cry, Consolability (FLACC ) Behavioral Pain Assessment Scale | Throughout the procedure of local anesthesia administration (which is approximately 8 minutes long), FLACC Scale was recorded by two trained and calibrated investigators independently.
  Face, Legs, Activity, Cry, Consolability (FLACC ) Behavioral Pain Assessment Scale scores range from 0 to 10 where higher scores indicate more severe pain and discomfort.

SECONDARY OUTCOMES:
Heart Rate(HR) | HR was recorded 5 times: 1) once subject is on the dental chair; 2) video on (about 3 min later); 3) topical anesthesia (about 2 min later); 4) needle insertion (about 2 min later); 5) immediately after local anesthesia is complete (about 1 min later).
  Heart beats per minute measured using a pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Osama M Felemban, BDS, DScD, Principal Investigator — King Abdulaziz University
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Felemban OM, Alshamrani RM, Aljeddawi DH, Bagher SM. Effect of virtual reality distraction on pain and anxiety during infiltration anesthesia in pediatric patients: a randomized clinical trial. BMC Oral Health. 2021 Jun 25;21(1):321. doi: 10.1186/s12903-021-01678-x. PMID 34172032